CLINICAL TRIAL: NCT01483196
Title: Feasibility Study of Vascular and Cognitive Assessments During Adjuvant Chemotherapy for Breast Cancer (VASCOG)
Brief Title: Vascular and Cognitive Assessments in Patients With Breast Cancer Undergoing Chemotherapy After Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB00017948; NCI-2011-02361 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CCCWFU 74111 (Other: Wake Forest University Health Sciences)
Record Dates: First submitted 2011-10-21; First posted 2011-12-01 (Estimated); Last update posted 2018-07-03 (Actual); Status verified 2018-07

CONDITIONS: Cognitive/Functional Effects; Recurrent Breast Cancer; Stage IA Breast Cancer; Stage IB Breast Cancer; Stage II Breast Cancer; Stage IIIA Breast Cancer; Stage IIIB Breast Cancer; Stage IIIC Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — High-Energy Shock Waves; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Diagnostic (TCD) (Experimental): Patients undergo TCD examination including bilateral evaluation of standard intracranial arterial segments including the M1 and M2 segments of the MCA, the ACA and PCA, via the transtemporal acoustic windows, the ICA siphon via transorbital approach, and the vertebral and basilar arteries (proximal, mid, and distal) via the suboccipital approach. Patients also undergo MRI. All tests occur between 21 days after completion of surgery and up to 30 days prior to adjuvant chemotherapy and between 20-60 days after completion of adjuvant chemotherapy.
  Interventions: Procedure: ultrasound imaging; Other: questionnaire administration; Procedure: assessment of therapy complications; Procedure: quality-of-life assessment; Procedure: magnetic resonance imaging

INTERVENTIONS:
Procedure: ultrasound imaging — Undergo TCD
  Other Names: ultrasonography; ultrasound; ultrasound test
Other: questionnaire administration — Complete neurocognitive questionnaires
Procedure: assessment of therapy complications — Undergo TCD
Procedure: quality-of-life assessment — Ancillary studies
  Other Names: quality of life assessment
Procedure: magnetic resonance imaging — Undergo MRI
  Other Names: MRI; NMR imaging; NMRI; nuclear magnetic resonance imaging

SUMMARY:
This clinical trial studies vascular and cognitive assessments in patients with breast cancer undergoing chemotherapy after surgery. Learning about vascular and cognitive function may help plan treatment and improve the quality of life of breast cancer patients. Transcranial Doppler ultrasound (TCD) may help study the side effects of chemotherapy in breast cancer patients and allow doctors to plan better treatment

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the feasibility of enrolling women who are receiving adjuvant chemotherapy for breast cancer to a clinical trial with assessments of vascular function and cognition before and after adjuvant chemotherapy and to obtain pilot data on outcomes that will be used in future larger-scale trials.

SECONDARY OBJECTIVES:

I. Evaluate the presence, duration, and severity of brain circulation changes identified with transcranial Doppler ultrasound (TCD) after adjuvant chemotherapy for breast cancer.

II. Assess the changes in flow-mediated dilation (FMD) and aortic dilation that occur after adjuvant chemotherapy for breast cancer.

III. Assess for correlation between the presence of brain circulation and vascular changes and performance on neuropsychological testing and the Functional Assessment of Cancer Therapy-Cognitive Scale (FACT-Cog).

OUTLINE:

Patients undergo TCD examination including bilateral evaluation of standard intracranial arterial segments including the M1 and M2 segments of the middle cerebral artery (MCA), the anterior cerebral artery (ACA) and posterior (PCA) cerebral artery, via the transtemporal acoustic windows, the internal carotid artery (ICA) siphon via transorbital approach, and the vertebral and basilar arteries (proximal, mid, and distal) via the suboccipital approach. Patients also undergo magnetic resonance imaging (MRI). All tests occur between 21 days after completion of surgery and up to 30 days prior to adjuvant chemotherapy and between 20-60 days after completion of adjuvant chemotherapy.

After completion of study treatment, patients are followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed non-metastatic breast cancer; stages 1-3 are acceptable
* Patients must be candidates for either neoadjuvant or adjuvant chemotherapy for breast cancer
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who have had prior systemic chemotherapy are not eligible for the study
* Patients who are scheduled to receive trastuzumab and/or bevacizumab are not eligible
* Patients who are on dialysis
* Women who are pregnant are not eligible due to unknown risks and potential harm to the unborn fetus
* Patients with metastatic breast cancer are not eligible

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Participation rate | Over 1 year
  Defined as the proportion of patients who participate in the study divided by the number of eligible patients. An exact binomial confidence interval (CI) will be calculated for this estimate.
Retention rate | Over 1 year
  Defined as the proportion of participating patients who complete measurements pre and post chemotherapy. An exact CI will also be calculated for this estimate.

SECONDARY OUTCOMES:
Changes in flow-mediated dilation and aortic dilation that occur after adjuvant chemotherapy for breast cancer | Approximately 90 days
Correlation between the presence of brain circulation and vascular changes and performance on neuropsychological testing and the FACT-Cog | approximately 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Heidi Klepin, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States